CLINICAL TRIAL: NCT06035848
Title: Components of Metabolic Derangement and Paracentesis for Determination of Surgery in Preterm Neonates With Necrotizing Enterocolitis.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In June 2023, it was decided to perform an intermediate analysis to assess the benefit or harm of the intervention.
Sponsor: Gerardo Fernández Ortega (Other Government)
Collaborators: Instituto Materno Infantil del Estado de México (Unknown); Instituto de Salud del Estado de México (Unknown)
Responsible Party: Sponsor-Investigator, Gerardo Fernández Ortega, Pediatric Surgery Specialty Coordinator / Principal Investigator, Hospital General de Mexico
Organization: Hospital General de Mexico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-2021
Record Dates: First submitted 2023-07-04; First posted 2023-09-13 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Necrotizing Enterocolitis
Keywords: Surgery; New born; Pediatrics; Mortality
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Paracentesis

STUDY DESIGN:
Intervention Model Description: The aim of this study was to determine an indication for early surgery in preterm neonates with necrotizing enterocolitis by using paracentesis in combination with the components of metabolic derangement compared to using the Bell´s criteria.
  Two groups of patients were formed (Control and Intervention). Control group: determination of surgery in a conventional manner according to Bell's criteria (absolute indication: pneumoperitoneum), with radiographic surveillance every 6 hours.
  Intervention Group: components of metabolic derangement measurement every 3rd day, it was considered positive when 3 or more points were present. These patients underwent paracentesis and if it was positive (faecal aspiration, serous fluid with Gram + staining, or serohematic fluid) the decision for surgery was made.
Who Masked: Participant, Investigator
Masking Description: The diagnosis, application of randomization to each group and blood sampling were performed by the neonatology staff, both the patients and the surgical team that provided care were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Components of metabolic derangement measurement every 3rd day, it was considered positive when 3 or more points were present. These patients underwent paracentesis and if it was positive (faecal aspiration, serous fluid with Gram + staining, or serohematic fluid) the decision for surgery was made.
  Interventions: Procedure: Association of the components of metabolic derangement and paracentesis.
- Control group (Active Comparator): Determination of surgery in a conventional manner according to Bell's criteria (absolute indication: pneumoperitoneum), with radiographic surveillance every 6 hours.
  Interventions: Procedure: Bell's criteria: pneumoperitoneum

INTERVENTIONS:
Procedure: Association of the components of metabolic derangement and paracentesis. — In the intervention group were determined:
  1. Components of metabolic derangement
  2. Paracentesis. Determination of surgery: 3 positive points of the components of the metabolic derangement and a positive paracentesis.
  The components of the metabolic derangement are the 7 parameters described by Tepas: positive blood culture, metabolic acidosis, neutropenia, bandemia, thrombocytopenia, hyponatremia and hypotension, being considered positive when 3 or more parameters are present.
  Paracentesis was considered positive according to Kosloske's criteria: obtaining more than 0.5ml of serohematic fluid, Gram-positive fluid and obtaining fecal material.
  Both groups had the same pre, trans and postoperative care.
  Other Names: MD7: components of metabolic derangement
  Arms: Intervention group
Procedure: Bell's criteria: pneumoperitoneum — In the control group, the surgery was determined according to Bell's criteria, in the presence of radiographic pneumoperitoneum as an absolute indication for surgery.
  Arms: Control group

SUMMARY:
The aim of this clinical trial is to associate paracentesis with positive metabolic derangement components for surgical determination in preterm infants with necrotizing enterocolitis. The main questions it aims to answer are:

* are the combination of metabolic derangement components and paracentesis good indicators for determining early surgery in preterm patients with necrotizing enterocolitis?
* With the use of the previously mentioned indicators, can mortality in these patients be reduced? Participants will undergo determination of the 7 parameters of the metabolic deterioration components and those with three or more positive points will undergo paracentesis and if this is also positive, it will be determined that the patient requires surgical management.

The researchers will compare with a control group to see the differences in surgical variables (length of necrotic bowel, length of viable bowel, need for intestinal diversion and surgical reintervention) and mortality.

DETAILED DESCRIPTION:
Controlled, randomized, double-blind clinical trial approved by the hospital's Ethics and Research Committee, subject to the Declaration of Helsinki. This study follows the CONSORT trial reporting guidelines. Patients younger than 37 weeks of gestation, with NEC stage IIa or greater according to Bell criteria were included.

Two groups of patients were formed (Control and Intervention), randomization was based on a randomization sequence generated using the Graphard 2021 program.

Control group: determination of surgery in a conventional manner according to Bell's criteria (absolute indication: pneumoperitoneum), with radiographic surveillance every 6 hours.

Intervention Group: CMD measurement every 3rd day, it was considered positive when 3 or more points were present. These patients underwent paracentesis and if it was positive (faecal aspiration, serous fluid with Gram + staining, or serohematic fluid) the decision for surgery was made.

Both groups received the same pre- and post-surgical medical management by neonatology.

As a safety criterion, it was defined that when a surgeon considered that a neonate had an indication for surgery, in spite of not meeting the criteria previously indicated for each group, the surgical intervention would be performed.

The diagnosis, implementation of the randomization to each group, and blood sampling were performed by the neonatology staff, the surgical research team being blinded; paracentesis was performed by a pediatric surgeon in the patient's crib with asepsis measures, antisepsis with chlorhexidine, sedation and analgesia (fentanyl 2 to 4 mcg /kg/dose), 1% lidocaine infiltration at the puncture site (iliac fossa right), a 22 G punzocath and a 10 ml syringe were used .

Follow-up was performed until the patient was discharged or died. Mortality was the dependent variable. The time from the patient's admission to the study until surgery was considered; during exploratory laparotomy, the length of intestinal necrosis, length of viable intestine, need for intestinal bypass, surgical intervention performed, and surgical reintervention were determined. In addition, fasting days and parenteral nutrition (TPN) were quantified.

Sample size. Based on the calculation for the difference of two proportions, a size of 31 patients per group was obtained, with a mortality difference of 30%, one-tailed, alpha of 5%, and statistical power of 80%. In June 2022, it was decided to carry out an intermediate analysis to assess the benefit or harm of the intervention, determined by the p value ˂ 0.05 in the dependent variable.

Statistical analysis. Descriptive statistics with measures of central tendency and dispersion were used. For qualitative variables frequencies and percentages, for quantitative variables mean and standard deviation. The Shapiro-Wilk test was used to test normal distribution.

For inferential statistics, group comparisons were performed using the χ2 test, Fisher's exact test, Student's t test or Mann Whitney U test, according to the type and distribution of the variable. The relative risk (RR) was obtained as a measure of association, with 95% confidence interval (CI). In addition, a bivariate analysis was performed between mortality and secondary variables. Statistical significance was established with a p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients equal to or less than 36.6 weeks gestation, with a diagnosis of NEC stage II A or greater according to Bell criteria.

Exclusion Criteria:

* Patients with a history of gastroschisis, suspected Hirschsprung's disease. Patients who do not give authorization for participation.

Elimination criteria:

Patients who during follow-up died due to some other condition. Patients who during the study declined to participate. Patients who in the surgical findings had data of Spontaneous Intestinal Perforation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality in preterm newborns with necrotizing enterocolitis | Neonates were followed from the date of surgery until death or hospital discharge, whichever came first, evaluated up to 6 months.
  The mortality of patients with necrotizing enterocolitis who required surgical management in both groups was determined.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Fernández, MD, Principal Investigator — Not affiliated
Locations (1):
- Hospital de Ginecología y Obstetricia IMIEM, Toluca, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez Ortega G, Martin De Saro MD, Cuevas Covarrubias SA, Moron Garcia GC, Plaza Benhumea L. Surgical decision-making strategies in preterm neonates with necrotizing enterocolitis: A randomized controlled clinical trial. Cir Pediatr. 2026 Jan 15;39(1):15-21. doi: 10.54847/cp.2026.01.13. English, Spanish. PMID 41550050